CLINICAL TRIAL: NCT04575441
Title: The Effects of Exercises With Pilates Ball on Balance, Reaction Time and Dual-task Performance of Kindergarten Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eastern Mediterranean University (Other)
Responsible Party: Principal Investigator, Zehra Güçhan, Dr., Eastern Mediterranean University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2019/0211
Record Dates: First submitted 2020-09-27; First posted 2020-10-05 (Actual); Last update posted 2020-12-03 (Actual); Status verified 2020-12

CONDITIONS: Healthy
Keywords: preschool children; physical fitness; exercise; physical activity
MeSH Terms: conditions — Motor Activity | interventions — Exercise

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pilates Ball Exercises (Experimental): Various exercises are conducted with using pilates ball. Sensory feedbacks like proprioception and vestibulation are given. Many physical fitness parameters like balance, coordination, speed and agility are used in this exercise program. Children are taken to the program for 40 min, twice a week during 6 weeks.
  Interventions: Other: Exercise with pilates ball
- Without exercise (No Intervention): The children in this group are not included in any kind of exercise/sport program during 6 weeks.

INTERVENTIONS:
Other: Exercise with pilates ball — Pilates ball exercises are used to give various sensory stimulation and increase motor skills. Children usually enjoy these kind of exercises as there is ball in every movement.
  Arms: Pilates Ball Exercises

SUMMARY:
The aim of this study is to investigate the effects of exercises conducted with pilates ball on balance, reaction time, quality of life, and behavior among preschool children.

60 volunteers, aged 4 and 5 years old, who continue kindergartens will randomly be grouped into two as study group (SG) (n=30) and control group (CG) (n=30). Exercises including pilates ball will be applied to SG children for 40 minutes, twice a week, 6 weeks. CG will continue normal daily routines for 6 weeks.

Sociodemographic information of all people will be recorded after their parents signed informed consent form. Single Leg Standing (eyes open and close) for static balance, Functional Reach Test (FRT)for dynamic balance, Ruler Drop Test for reaction time, dual task performance methods will be used.

DETAILED DESCRIPTION:
Exercises are generally suggested starting from primary school children. However, exercise habit should be given to people from earlier ages. Moreover, doing exercise can be beneficial to improve motor skills of this age and this improvement can support other developmental areas of these children. Thus, this study aims to investigate the effects of an exercise routine on balance, reaction time and dual task performance of preschool children. This exercise program includes pilates ball to make more fun for this age group. All movements are conducted with the same pilates ball. Exercises are conducted with individual sessions in the kindergartens of children.

ELIGIBILITY:
Inclusion Criteria:

* having a birth year 2015 or 2016.

Exclusion Criteria:

* Having cognitive, physical and/or orthopedic problem
* Any pain which may prevent doing exercise
* Having visual and/or auditory loss

Ages: 4 Years to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 62 (Actual)
Dates: Start 2020-05-01 (Actual); Primary Completion 2020-10-01 (Actual); Study Completion 2020-10-10 (Actual)

PRIMARY OUTCOMES:
Dynamic balance | change from baseline at 6 weeks
  Functional reach test is used. Children are asked to stand next to the wall with their right side and extend their right arm with 90 degree shoulder flexion. Then they are asked to extend with their arm as far as possible by protecting their lower limb posture. The distance is recorded in cm.

SECONDARY OUTCOMES:
Static balance | change from baseline at 6 weeks
  Children are asked to stand on dominant leg. Their standing duration is recorded.
Reaction time | change from baseline at 6 weeks
  Ruler drop test is used to measure reaction time. A rule of 50 cm long is used. Children are asked to catch the ruler as fast as possible. Since the ruler is left with its zero point below, distance is recorded in cm as the result of this outcome.
Dual task performance | change from baseline at 6 weeks
  Timed-up and go (TUG) test is used as a motor skill and a cognitive task is asked from children as a second task. For timed up and go test, a three meter pathway will be marked with red colored masking tape. The TUG test is administered using 2 standard chairs and children are asked to walk in a self preferred speed. At the same time, children are asked to count many animal names.

CONTACTS AND LOCATIONS:
Overall Officials: Zehra Güçhan Topcu, Dr., Study Director — Eastern Mediterranean University
Locations (1):
- Zehra Güçhan Topcu, Famagusta, Cyprus

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Obuz T, Topcu ZG. The effects of exercises with a Pilates ball on balance, reaction time and dual-task performance of kindergarten children. J Comp Eff Res. 2022 Jun;11(8):583-593. doi: 10.2217/cer-2021-0293. Epub 2022 May 6. PMID 35514277